CLINICAL TRIAL: NCT05321251
Title: Topical Insulin Drops for the Treatment of Neurotrophic Keratopathy.
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study never commenced due to logistical issues.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00107280
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Neurotrophic Keratitis
Keywords: topical insulin; neurotrophic keratopathy; neurotrophic keratitis; tarsorrhaphy
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial for the treatment of neurotrophic keratitis. Topical insulin drops will be compared to the current gold standard treatment temporary tarsorrhaphy. Patients will be recruited in Vancouver, Edmonton, Toronto, Montreal, and Halifax. Patients with neurotrophic corneal ulcers will be identified through the Ophthalmology on call resident clinics in each location. They will be directly referred to a physician in their city who is participating in this study. At least 12 patients will be enrolled in each group (as per power calculation): topical insulin drops or tarsorrhaphy.
Masking Description: Treatment will be randomized / assigned randomly, but neither the patients, care providers, or investigators will be masked to treatment once it is being provided.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical insulin (Experimental): Topical insulin (Humulin R) will be compounded under sterile conditions at a local pharmacy at a concentration of 25 IU / ml in sterile balanced saline solution (0.9%). Topical insulin will be administered four times per day to the affected eye. A bottle of topical insulin can be used for 14 days. Any remaining topical insulin will be discarded as waste after 14 days.
  Interventions: Drug: Insulin
- Tarsorrhaphy (Active Comparator): Patients in this group will receive a temporary, central tarsorrhaphy and will not use additional eye drops.
  Interventions: Procedure: Tarsorrhaphy

INTERVENTIONS:
Drug: Insulin — see arm description
  Arms: Topical insulin
Procedure: Tarsorrhaphy — see arm description
  Arms: Tarsorrhaphy

SUMMARY:
Many diseases can affect corneal nerves. Corneas that lack normal sensation are considered neurotrophic. Neurotrophic corneas are predisposed to persistent epithelial defects, recurrent erosions, and corneal ulcers. These can lead to a variety of complications, from subjective pain, discomfort, and blurry vision, to corneal perforation and endophthalmitis. Neurotrophic corneas and the persistent epithelial defects associated with them can be very difficult to treat. Non-invasive measures include topical drops (artificial tears, antibiotics, or steroids), bandage contact lens, and punctal plugs. More invasive surgical treatments include membrane grafts, tarsorrhaphy, and keratoplasty. Despite these treatments, many neurotrophic corneas still do not heal. This study aims to test the efficacy of topical insulin in the treatment of neurotrophic keratopathy.

DETAILED DESCRIPTION:
Purpose: To trial topical insulin drops to promote healing in neurotrophic keratitis that has been refractory to conventional management versus tarsorrhaphy.

Hypothesis: Topical insulin might promote re-epithelialization in the setting of neurotrophic keratitis (Stage 2 or 3) with persistent epithelial defect refractory to conventional treatments and be a non-inferior treatment to tarsorrhaphy.

Justification: Several experiments support the use of insulin for the promotion of corneal epithelial healing. In vitro experiments with immortalized corneal epithelial cells suggest that insulin improves epithelial cell migration. A rabbit model showed improvement in corneal hypoesthesia after topical insulin exposure. These results suggest that early hypoesthesia may be reversible, and thereby improve epithelial wound healing. Another rabbit model showed that topical insulin might alter the corneal surface by increasing the tensile strength of corneal wounds. Finally, the presence of insulin receptors on the cornea and lacrimal gland suggests that insulin may contribute to corneal wound healing.

Few case studies describe the use of topical insulin in the absence of other concurrent treatments for neurotrophic keratitis.

Objectives: Through use of topical insulin, promotion of corneal healing in cases where conventional methods have failed. These include topical antibiotics, preservative free artificial tears, and bandage contact lens for at least 2 weeks. This study will evaluate topical insulin as a salvage treatment in patients who otherwise would require tarsorrhaphy.

Research Method: Patients will be recruited in Vancouver, Edmonton, Toronto, Ottawa, Halifax, and Montreal. Patients with neurotrophic corneal ulcers will be identified through the Ophthalmology on call resident clinics in each location and directly referred to a physician in their city who is participating in this study. At least 12 patients will be enrolled in each group (as per power calculation).

Baseline demographic information will be collected (age, gender, medical comorbidities, ocular comorbidities, current medications, and previous and current eyedrops). Baseline ocular examination will consist of a complete ophthalmologic exam, including visual acuity, intraocular pressure, dilated fundus exam or BScan imaging, corneal sensation, eyelid measurements (palpebral fissure, presence of entropion or ectropion, and lagophthalmos), and anterior segment exam and photography. Corneal sensation will be measured in group quadrants and centrally and quantified with cochet bonnet esthesiometry.

Patients will be randomized to one of two groups: Permanent medial tarsorrhaphy or topical insulin drops.

Patients will stop all other topical medication before commencing use of insulin eyedrops. Topical insulin will be compounded under sterile conditions at a local pharmacy at a concentration of 25 IU / ml in sterile balanced saline solution (0.9%). Topical insulin will be administered four times per day to the affected eye.

Patients will be followed up every 3 days after initiation of therapy, or as needed. Each follow up visit will include an ophthalmologic exam with repeat measurements of the epithelial defect, visual acuity, IOP, and anterior segment exam.

The primary outcome will be time to re-epithelialization of neurotrophic ulcer, defined as <0.5mm of remaining epithelial defect. There will also be an evaluation of the percentage of patients healed at each follow up time point. Subgroup analysis will analyze time to re-epithelialization in patients with diabetes separate from patients without diabetes.

The trial will be terminated early if the patients should develop adverse side effects, including allergy, worsening of symptoms, infection, or worsening of keratitis.

Plan for Data Analysis: Statistical analysis to determine the rate of improvement of neurotrophic keratitis by photograph analysis, corneal sensation in four quadrants and centrally, and visual acuity testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neurotrophic keratitis with persistent epithelial defect that has been refractory to conventional treatments for at least 2 weeks
* 18 years or older
* Able to provide informed consent
* Failed other conventional treatments for neurotrophic keratitis
* Understanding and accepting of use of topical insulin alone

Exclusion Criteria:

* Less than 18 years old
* Pregnant or breastfeeding women
* Unable to provide informed consent
* Unable to comply with tests/follow-up
* Lid function abnormalities (e.g., lagophthalmos, entropion, ectropion, or abnormal orbicularis function from cranial nerve 7 palsy or Bell's palsy)
* Patients who require ongoing topical treatment (e.g. topical ganciclovir)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Time to re-epithelialization of neurotrophic ulcer | 3 months
  Time taken for re-epithelialization of the neurotrophic ulcer which will be defined as <0.5 mm of the remaining epithelial defect

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Rudnisky, MD MPH, Principal Investigator — University of Alberta
Locations (6):
- Canada (6):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - Precision Cornea Clinic, Ottawa, Ontario
  - University of Toronto, Toronto, Ontario
  - University of Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galvis V, Nino CA, Tello A, Grice JM, Gomez MA. Topical insulin in neurotrophic keratopathy after resection of acoustic neuroma. Arch Soc Esp Oftalmol (Engl Ed). 2019 Feb;94(2):100-104. doi: 10.1016/j.oftal.2018.06.003. Epub 2018 Jul 17. English, Spanish. PMID 30025986
- [Background] Bastion ML, Ling KP. Topical insulin for healing of diabetic epithelial defects?: A retrospective review of corneal debridement during vitreoretinal surgery in Malaysian patients. Med J Malaysia. 2013 Jun;68(3):208-16. PMID 23749008
- [Background] Fai S, Ahem A, Mustapha M, Mohd Noh UK, Bastion MC. Randomized Controlled Trial of Topical Insulin for Healing Corneal Epithelial Defects Induced During Vitreoretinal Surgery in Diabetics. Asia Pac J Ophthalmol (Phila). 2017 Sep-Oct;6(5):418-424. doi: 10.22608/APO.201780. Epub 2017 Aug 22. PMID 28828764
- [Background] Tong CM, Iovieno A, Yeung SN. Topical insulin for neurotrophic corneal ulcers. Can J Ophthalmol. 2020 Oct;55(5):e170-e172. doi: 10.1016/j.jcjo.2020.04.001. Epub 2020 May 13. No abstract available. PMID 32416928
- [Background] Diaz-Valle D, Burgos-Blasco B, Gegundez-Fernandez JA, Garcia-Caride S, Puebla-Garcia V, Pena-Urbina P, Benitez-Del-Castillo JM. Topical insulin for refractory persistent corneal epithelial defects. Eur J Ophthalmol. 2021 Sep;31(5):2280-2286. doi: 10.1177/1120672120958307. Epub 2020 Sep 21. PMID 32951459
- [Result] Wang AL, Weinlander E, Metcalf BM, Barney NP, Gamm DM, Nehls SM, Struck MC. Use of Topical Insulin to Treat Refractory Neurotrophic Corneal Ulcers. Cornea. 2017 Nov;36(11):1426-1428. doi: 10.1097/ICO.0000000000001297. PMID 28742619